CLINICAL TRIAL: NCT03002376
Title: An Exploratory Tumor Biopsy-driven Study to Understand the Relationship Between Biomarkers and Indicators of Clinical Response in Immunomodulatory Treatment-naïve Unresectable Stage III/IV Melanoma Patients Receiving REGN2810 (Anti-PD-1)
Brief Title: An Exploratory Tumor Biopsy-driven Study to Understand the Relationship Between Biomarkers and Clinical Response in Melanoma Patients Receiving REGN2810 (Anti-PD-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1606; 2016-002755-16 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGN2810 (Experimental): REGN2810 treatment
  Interventions: Drug: REGN2810

INTERVENTIONS:
Drug: REGN2810 — REGN2810 treatment
  Other Names: cemiplimab; Libtayo

SUMMARY:
This study is being conducted to compare the relationship of patient response to treatment to changes in tumor environment.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of stage III (unresectable) or stage IV cutaneous melanoma (non-acral lentiginous) with at least 1 lesion that is measurable by RECIST 1.1 criteria and accessible for biopsies
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate hepatic function
* Adequate renal function
* Adequate bone marrow function
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent
* Able to understand and complete study-related questionnaires
* Anticipated life expectancy >12 weeks

Key Exclusion Criteria:

* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs).
* Prior treatment with an agent that blocks the programmed death-1/ programmed death-ligand 1 (PD-1/PD-L1 pathway)
* Prior treatment with other immune modulating anti-cancer agents, except for remote treatment (>6 months) in adjuvant setting.
* Untreated or active brain metastases or spinal cord compression
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of REGN2810

Other protocol-defined inclusion/exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in the tumor microenvironment and the change in tumor volume following REGN2810 treatment versus baseline | Baseline up to week 24

SECONDARY OUTCOMES:
Correlation between baseline tumor characteristics and the change in tumor volume following treatment in REGN2810 | Baseline up to week 24
Incidence of Adverse Event (AEs) in patients treated with REGN2810 | Baseline through treatment with REGN2810 (up to 48 weeks) and follow up
REGN2810 serum concentrations | Baseline up to 6 weeks following last dose of REGN2810
Anti-REGN2810 antibody levels | Baseline up to 6 weeks following last dose of REGN2810
The progression-free survival (PFS) in patients treated with REGN2810 | Baseline up to 6 weeks following last dose of REGN2810
The overall response rate in patients treated with REGN2810 | Baseline up to 6 weeks following last dose of REGN2810

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- Radboud University Medical Center, Nijmegen, Netherlands
- Military Medical Academy, Belgrade, Serbia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital-Yonsei University College of Medicine, Seoul
- United Kingdom (2):
  - Guy's Hospital and St. Thomas NHS Foundation Trust, London
  - Churchill Hospital, Oxford